CLINICAL TRIAL: NCT05770076
Title: Effect of Probiotic Lysate (Postbiotic and Metabiotic) Supplementation on Metabolic Parameters in Type 2 Diabetes Patients
Brief Title: Probiotic Lysate (Postbiotic and Metabiotic) Supplementation for Type 2 Diabetes Patients (DELI_Diab Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Collaborators: Taras Shevchenko National University of Kyiv (Other); Danylo Halytsky Lviv National Medical University (Other); Center for Innovative Medical Technologies of the National Academy of Sciences of Ukraine (Other); Kyiv City Clinical Endocrinology Center (Other); MirImmunoFarm (Unknown); Stellar Biotics (Unknown)
Responsible Party: Principal Investigator, Nazarii Kobyliak, Associate Professor, Endocrinology Department, Bogomolets National Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DELI_Diab
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Obesity; Obesity, Abdominal; Insulin Resistance; Insulin Sensitivity; Type2 Diabetes; Type 2 Diabetes Mellitus in Obese
Keywords: Postbiotics; metabiotics; L. rhamnosus; L. delbrueckii; Obesity; Type2 Diabetes; Insulin Resistance
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization was done by the study statistician based on a computer-generated list. The groups were homogeneous according to age, sex and diagnostic criteria. The assignment of groups was blind to participants, research staff and outcome assessors moreover, to maintain blind parallel study the statistician was not aware of the allocation of participants to intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic lysate (postbiotic and metabiotic) group (Active Comparator): oral, 2 capsules per day (BID) for 3 month treatment
  Interventions: Dietary Supplement: Probiotic lysate (postbiotic and metabiotic)
- Placebo group (Placebo Comparator): placebo, oral, 2 capsules per day (BID) for 3 month treatment
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic lysate (postbiotic and metabiotic) — Each capsule contains 100 mg of cell lysate and DNA fragments of the probiotic strain L. rhamnosus DV - NRRLB-68023 in powder
  Other Names: Del-Immune V® Extra
  Arms: Probiotic lysate (postbiotic and metabiotic) group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
The current study aim was to conduct placebo-controlled randomize clinical trial to assess the short-term efficacy and safety of postbiotics as an adjunction to the standard anti-diabetic therapy on insulin resistance, glycemic control parameters, β-cells functional activity, anthropometric parameters and markers of a chronic systemic inflammatory response in type 2 diabetes patients.

The study will include 3 periods. Screening period of up to 1 weeks to assess the eligibility to inclusion/exclusion criteria. Treatment period for 3 month where the participants will receive a twice daily oral dose of postbiotics (cell lysate and DNA fragments of the probiotic strain L. rhamnosus DV - NRRLB-68023) at the assigned dose of 100mg or placebo in capsules. During this period monthly phone contacts will be done for assessment of compliance and safety concerns. Follow-up period of up to 3 month.

DETAILED DESCRIPTION:
The scientific literature points to the beneficial properties of probiotics in the process of regulating metabolism, yet at the same time, some scientific papers question the effectiveness and the safety of probiotics. In turn, postbiotics and metabiotics are preparations of inanimate microorganisms and / or their components, which are directly identified with the safety of their use and the health benefits of the host. Due to the chemical structure of postbiotics and metabiotics, it is found that they have many health benefits; in particular, they have a local effect on certain tissues of the intestinal epithelium, and influence on many other organs and tissues. It is postbiotics metabolites and metabiotics structural cell fragments that create the appearance of a therapeutic effect of probiotics, which, in turn, limits the risk of introducing living microorganisms into a weakened immune defence. It should also be pointed out that postbiotics and metabiotics are more stable and have a longer shelf-life.

The practical use of probiotics and the study of the mechanism of their action made lately to find that a certain level of biological activity is preserved by dead probiotic cells and even their lysates, which are the natural mixes of metabiotic and postbiotic substances; a biological activity which is strongly oriented toward gut health and immune system regulation. Because probiotic lysates demonstrated biological activity without any of the potential adverse side effects associated with live bacterial cells, one of the future goal is research of the novel postbiotics and metabiotics substances, their individual structures and biological characteristics for understanding their way of communications with host cells and microbiota representatives.

Considering the high biological activity and safety of postbiotics and metabiotic substances, it can be concluded that such a treatment vector will be promising in the near future. That's why our investigation will concentrate on postbiotic, a supplement containing dry fermented cell lysate and DNA fragments of the probiotic strain L. rhamnosus DV - NRRLB-68023.

Recent scientific animal studies on the stated issues point to the benefits of some postbiotics in treating metabolic disorders. The current study aim was to conduct placebo-controlled randomize clinical trial to assess the short-term efficacy and safety of postbiotics as an adjunction to the standard anti-diabetic therapy on insulin resistance, glycemic control parameters, β-cells functional activity, anthropometric parameters and markers of a chronic systemic inflammatory response in type 2 diabetes patients.

The study will include 3 periods. Screening period of up to 1 weeks to assess the eligibility to inclusion/exclusion criteria. Treatment period for 3 month where the participants will receive a twice daily oral dose of postbiotics (cell lysate and DNA fragments of the probiotic strain L. rhamnosus DV - NRRLB-68023) at the assigned dose of 100mg or placebo in capsules. All capsules will be identical with similar organoleptic characteristics (e.g., taste and appearance).. Follow-up period of up to 3 month.

The pre-randomization period will be designed to minimize the effects of dietary changes on metabolic markers. For this purpose, 2 weeks before the study start, after inform consent signed, patients were instructed in one-on-one sessions with a dietitian to follow a therapeutic lifestyle-change diet as classiﬁed by the NCEP. In addition, participants were instructed to continue with stable anti-hyperglycemic treatment and received standardized mild physical training for 1 hour per day.

Patients who underwent the study were instructed to take the trial medication as prescribed. Throughout the study, weekly phone follow-up visits were provided for assessment of compliance, adherence to the protocol, as well as the recording of adverse events. The effectiveness of therapy was compared and evaluated separately in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* adult participants (ages 18-70)
* presence of T2D diagnosed according to criteria of the American Diabetes Association;
* BMI 25-40 kg/m2;
* patient who treated with diet and exercise alone or metformin, SUs and insulin on a stabilized dose for at least 3 months before the study;
* daily insulin dosage less than 60IU;
* HbA1c between 6.5 and 10.0 %;
* written informed consent.

Exclusion Criteria:

* presence of type 1 diabetes;
* severe diabetes-related complications at screening (ie, end-stage DKD, neuropathy requiring pharmacological treatment, proliferative retinopathy, autonomic neuropathy);
* treatment with other than mention in inclusion criteria antidiabetic drugs (pioglitazone, SGLT-2 antagonists, GLP-1 analogues, DPP IV inhibitors etc);
* regular use of an agents with gut microbiota modulation activity (antibiotic, pro-, pre-, post or synbiotics supplement etc.) within 3 months prior to enrollment;
* allergy on probiotics or their components;
* presence of gastrointestinal diseases such as food allergy, celiac disease, non-specific ulcerative colitis;
* uncontrolled cardiovascular or respiratory disease, decompensated liver disease including ascites, encephalopathy or variceal bleeding, active malignancy, or chronic infections;
* participant who had severe course of COVID-19 (extracorporeal membrane oxygenation, mechanically ventilated), and/or had a confirmed case of COVID-19 within 4 weeks prior to enrollment;
* participation in other clinical trials;
* presence of pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1c level | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline
  HbA1c in %
Changes in fasting plasma glucose (FPG) level | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline
  FPG in mmol/L

SECONDARY OUTCOMES:
HOMA-2IR | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline
  This model can be calculated using the software supplied by the Oxford Centre for Diabetes Endocrinology and Metabolism available at http://www.dtu.ox.ac.uk/homacalculator/index.php
insulin sensitivity (%S) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline
  This model can be calculated using the software supplied by the Oxford Centre for Diabetes Endocrinology and Metabolism available at http://www.dtu.ox.ac.uk/homacalculator/index.php
  [Time Frame: 8 weeks compared to baseline]
β-cell function (%B) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline
  This model can be calculated using the software supplied by the Oxford Centre for Diabetes Endocrinology and Metabolism available at http://www.dtu.ox.ac.uk/homacalculator/index.php
  [Time Frame: 8 weeks compared to baseline]
C-peptide | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline
  C-peptide, ng/ml
High censitivity CRP (C-reactive Protein) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline
  hs-CRP in mg/L
weight | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline
  weight in kg
waist circumferences (WC) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline
  WC in cm
body mass index (BMI) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline
  weight in kg and height in meters will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Nazarii Kobyliak, PhD, Principal Investigator — Bogomolets National Medical University
Locations (4):
- Ukraine (4):
  - Bogomolets National Medical University, Kyiv
  - Kyiv City Clinical Endocrinology Center, Kyiv
  - Center for Innovative Medical Technologies of the National Academy of Sciences of Ukraine, Kyiv
  - Danylo Halytsky Lviv National Medical University, Lviv